CLINICAL TRIAL: NCT00502164
Title: A Phase I Open-label Dose Escalation Study to Assess the Safety and Tolerability of AZD2171 Following Multiple Oral Doses in Subjects With Advanced Prostate Cancer.
Brief Title: Study to Assess Safety and Tolerability of AZD2171 After Multiple Doses in Patients With Advanced Prostate Cancer
Acronym: AZD2171IL/0003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00003
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Prostate Adenocarcinoma
Keywords: Advanced Prostate Cancer
MeSH Terms: interventions — cediranib

INTERVENTIONS:
Drug: AZD2171

SUMMARY:
A study to assess safety and tolerability of AZD2171 after multiple doses in patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men, 18yrs and older
* Histological or cytological confirmation of prostate adenocarcinoma (symptomatic or asymptomatic)
* Prior hormonal therapy, and/or no more than 1 prior chemotherapy regimen (including estramustine and/or corticosteroids) for treatment of prostate adenocarcinoma

Exclusion Criteria:

* Prior radiotherapy to bone metastases within 4 weeks prior to screening
* any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy
* Brain metastases or spinal cord compression, unless treated at least 4 weeks before entry, and stable with steroid treatment for 1 week.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-03

PRIMARY OUTCOMES:
To establish the safety and tolerability of AZD2171 in subjects with advanced prostate adenocarcinoma

SECONDARY OUTCOMES:
Explore the PK profile of AZD2171 at steady-state administration to subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nick Botwood, BSc, MBBS, MRCP, MFPM, Study Director — AstraZeneca; Eric Small, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - Research Site, Nashville, Tennessee